CLINICAL TRIAL: NCT05887128
Title: Accuracy of Extra-oral Bite-wing Radiography in Detecting Calculus and Crestal Bone Loss
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 22-2079
Record Dates: First submitted 2023-02-21; First posted 2023-06-02 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Periodontitis; Calculus, Dental; Bone Loss, Alveolar
MeSH Terms: conditions — Periodontitis; Dental Calculus; Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To compare the diagnostic accuracy of extra-oral x-rays with intra-oral x-rays, in contrast to clinically observed measurements, for the detection of calculus and bone loss of either the suprabony or infrabony types in patients undergoing periodontal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be active patients of record at CU School of Dental Medicine
* Patients will have an active treatment plan for periodontal open flap surgery
* Patients will be classified as either ASA I or ASA II
* Patients must have periodontal probing depths >/= 5mm and radiographic sings of marginal bone loss (supra or infra bony)

Exclusion Criteria:

* Less than 18 years of age
* ASA III or above
* Emergency patients
* Pregnant patients
* Patients who are not patients of record at the CU School of Dental Medicine
* Patients with a recent panoramic radiograph that contraindicates the need for new imaging in the form of extra-oral bitewings

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 40 individuals who are currently active patients at the University of Colorado School of Dental Medicine Graduate Periodontics Department. Intra-oral x-rays will be taken on examination, which is the standard of care. Patients who require periodontal surgery and have signed treatment plans to undergo the surgery will be asked to participate in the study. Extra-oral x-rays will be taken at that time, which is for research purpose. This is the same exposure as a panoramic x-ray, which is the standard of care to receive along with the intra-oral x-rays. Patients will be excluded if they have a recent panoramic x-ray.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic evidence of calculus | Baseline - Yes or No
  Radiographic evidence of calculus
Radiographic measure of alveolar bone loss | Baseline - measured in mm
  Radiographic measure (mm) of alveolar bone loss, as measured from the Cemento-enamel-junction to base of defect
Clinical evidence of calculus | Baseline - Yes or No
  Clinical evidence of calculus
Clinical measure of alveolar bone loss | Baseline - measured in mm
  Clinical measure (mm) of alveolar bone loss, as measured from Cemento-enamel-junction to base of defect using a periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: William Carter, DDS, Principal Investigator — University of Colorado, Denver
Locations (1):
- Univeristy of Colorado School of Dental Medicine Dental Clinic, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No